CLINICAL TRIAL: NCT02028234
Title: "Pharmacodynamic Comparison of Omeprazole Versus Pantoprazole on Platelet Reactivity in Patients With Acute Coronary Syndromes on Dual Antiplatelet Therapy With New P2Y12 Inhibitors"
Brief Title: "Pharmacodynamic Comparison of Omeprazole Versus Pantoprazole on Platelet Reactivity in Patients With Acute Coronary Syndromes on Dual Antiplatelet Therapy With New P2Y12 Inhibitors" -Trial dOPPLER-
Acronym: dOPPLER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Polacco Marina, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010114
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Pantoprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pantoprazole (Active Comparator): Patients were randomly assigned to omeprazole (20 mg day) or pantoprazole (20 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Interventions: Drug: Pantoprazole,; Drug: Omeprazole
- Omeprazole (Active Comparator): Patients were randomly assigned to omeprazole (20 mg day) or pantoprazole (20 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Interventions: Drug: Pantoprazole,; Drug: Omeprazole

INTERVENTIONS:
Drug: Pantoprazole, — os, 20 mg, once per day, for 30 days
  Other Names: pantorc
Drug: Omeprazole — os, 20 mg, once per day, for 30 days
  Other Names: lansox

SUMMARY:
Clopidogrel and Prasugrel are pro-drug necessitating conversion in active metabolites through CYP 450 system (CYP), particularly CYP3A and CYP2C19 isoforms.

These drugs are platelet purinergic receptor antagonists, known as P2Y12. The link between active metabolite of Clopidogrel and Prasugrel to P2Y12 receptor prevents ADP receptor activation and inhibits several events leading to conformational change of platelets, therefore facilitating their activation and aggregation, that is the basis of acute coronary syndromes. Proton pump inhibitors (PPI) are actually considered principal agents reducing gastroenteric bleeding risk associated to antiplatelet therapy. Nevertheless the interaction between PPI and antiplatelet therapy has been object of interest. Several studies demonstrated PPI reduce efficacy of clopidogrel on platelet reactivity. Only few data about Prasugrel are available showing a minor effect of PPI on its antiplatelet activity than clopidogrel. Differing from prasugrel and clopidogrel, ticagrelor is a direct inhibitor of P2Y12, not necessitating biotransformation in the liver; therefore its interaction with PPI remains unclear. Interaction between omeprazole and clopidogrel seems related to high inhibitory activity of PPI on CYP2C19, interfering with the conversion of clopidogrel in its active metabolite.

DETAILED DESCRIPTION:
Clopidogrel and Prasugrel are pro-drug necessitating conversion in active metabolites through CYP 450 system (CYP), particularly CYP3A and CYP2C19 isoforms.

These drugs are platelet purinergic receptor antagonists, known as P2Y12. The link between active metabolite of Clopidogrel and Prasugrel to P2Y12 receptor prevents ADP receptor activation and inhibits several events leading to conformational change of platelets, therefore facilitating their activation and aggregation, that is the basis of acute coronary syndromes.

Despite double antiplatelet drugs are the principle therapy for the treatment and the prevention of atherothrombotic events in cardiovascular diseases, they are the most important cause of bleeding peptic ulcer. Proton pump inhibitors (PPI) are actually considered principal agents reducing gastroenteric bleeding risk associated to antiplatelet therapy. Nevertheless the interaction between PPI and antiplatelet therapy has been object of interest. Several studies demonstrated PPI reduce efficacy of clopidogrel on platelet reactivity, probably through the inhibition of its metabolism, increasing the risk of cardiovascular events. Only few data about Prasugrel are available showing a minor effect of PPI on its antiplatelet activity than clopidogrel. Differing from prasugrel and clopidogrel, ticagrelor is a direct inhibitor of P2Y12, not necessitating biotransformation in the liver; therefore its interaction with PPI remains unclear. Nevertheless actual studies considered only clinical outcomes (MACEs), such as a subgroup analysis of the Platelet Inhibition and Patient Outcomes (PLATO) trial, showing a higher rate of MACEs in clopidogrel and Ticagrelor patients undergone PPI therapy, especially omeprazole treatment. Interaction between omeprazole and clopidogrel seems related to high inhibitory activity of PPI on CYP2C19, interfering with the conversion of clopidogrel in its active metabolite. It is yet unclear the higher rate of MACEs in the ticagrelor group, similarly to clopidogrel, despite it hasn't a hepatic metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients undergone PTCA in our institution in the period between July 2013 and December 2013 will be eligible to be enrolled.
2. Positive biomarker indicating myocardial necrosis.
3. All patients with prior myocardial infarction (MI) or coronary artery bypass grafting; coronary artery disease will be included.

Exclusion Criteria:

1. Increased risk of bleeding (ex. active bleeding, major surgery <30 days).
2. Allergy or adverse reactions to administered drugs.
3. Other drugs or medications that affect CYP3A4 mediated drug metabolism.
4. Patients with missing follow-up data will be dropped out from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 30 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California]

SECONDARY OUTCOMES:
Frequency of high platelet reactivity | After 30 days of treatment with each drug
  Frequency of high platelet reactivity with the 2 study treatments (as defined by a Platelet Reaction Unit value>240

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza Univeristy of Rome, Rome, Italy, Italy